CLINICAL TRIAL: NCT04523402
Title: Oxaliplatin and Gemcitabine (GEMOX) Neoadjuvant Therapy for Resectable Intrahepatic Cholangiocarcinoma With High Risk of Lymph Node Metastasis as Preoperatively Evaluated by a Radiomics Model
Brief Title: Neoadjuvant Therapy for Resectable Intrahepatic Cholangiocarcinoma With High Predict Risk of Lymph Node Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Prof., Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2020-K-027
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Intrahepatic Cholangiocarcinoma Recurrent
Keywords: Intrahepatic Cholangiocarcinoma; Neoadjuvant chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemotherapy following liver section (Experimental): 1. GEMOX chemotherapy:
  1. It is performed within one week after the identification of ICC;
  2. Day1 Oxaliplatin 85mg/m2 + gemcitabine 1g/m2, Day 8 gemcitabine 1g/m2;
  3. Three weeks is a course of treatment;
  4. A total of 3 courses.
  2. Liver resection: It is performed 1 month after chemotherapy
  Interventions: Drug: Neoadjuvant chemotherapy
- Liver resection (No Intervention): Liver resection:
  It is performed within one week after the identification of ICC.

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Neoadjuvant chemotherapy with GEMOX regimen before liver resection
  Other Names: Preoperative chemotherapy
  Arms: Neoadjuvant chemotherapy following liver section

SUMMARY:
A randomized controlled, open label, phase II clinical trial is designed to target patients with resectable intrahepatic cholangiocarcinoma (ICC) with high risk of lymph node metastasis as evaluated by our previously established radiomics model, which has low postoperative recurrence-free survival. In this study, we aim to compare the prognosis of ICC patients who undergo liver resection (LR) following preoperative oxaliplatin and gemcitabine (GEMOX) neoadjuvant therapy (experimental arm) versus LR alone (control arm).

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) is the second most common liver cancer, and its incidence and mortality have been rising worldwide over the past two decades. Liver resection (LR) remains the only potentially curative treatment for ICC. However, the long-term outcome after LR is still dismal, and the 5-year survival after curative-intent resection was up to 35%. Lymph node (LN) metastasis is found in about 40% of ICC patients and is known to be one of the most important adverse prognostic factors. Considering such circumstances, it is crucial to determine the validity of routine LN dissection for ICC during LR, but there is so far no definitive evidence about the use of this surgical procedure. Preoperative individualized LN status assessment is beneficial for clinical decision of LN dissection and stratifying patients who may benefit from preoperative neoadjuvant therapy. The conventional and qualitative radiological characteristics in abdominal computerized tomography (CT) exhibited limited accuracy for preoperative assessment of LN status. Radiomics, a novel approach in medical image analysis, involves high-throughput extraction of quantitative image features and then associates these features with clinical concerns. The radiomic approach has been employed into preoperative diagnosis and prediction of prognosis. We have proposed a nomogram, incorporating conventional clinico-radiological characteristics and novel radiomic features in CT scan, provided accurate LN metastasis prediction in ICC patients and may aid the treatment decision making.

Neoadjuvant therapy refers to some treatments taken before surgery for newly treated tumor patients who have not found distant metastasis, including chemotherapy, radiotherapy, targeted therapy, etc., to reduce tumors, reduce tumor stages, and reduce postoperative recurrence rate, prolonging survival time. As suggested by the results from previous studies, neoadjuvant chemotherapy with oxaliplatin plus gemcitabine for locally advanced ICC may be an effective downstaging option, facilitating secondary resectability in patients with initially unresectable disease (53%, 39 in 74 patients received secondary resection). In addition, for selected patients with locally advanced ICC who showed pre-transplant disease stability on neoadjuvant chemotherapy could obtain 50% 5-year recurrence-free survival and 83.3% 5-year overall survival.

These evidences suggest that neoadjuvant chemotherapy with GEMOX regimen may be an ideal modality for patients with resectable ICC with high possibility of LN metastasis to reduce potential risk of recurrence, which is worth more investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent;
2. Male or female patients aged 18-70;
3. Eastern Cooperative Oncology Group (ECOG) score 0 points, Child-Pugh rating A;
4. Clinically diagnosed as ICC as a potential entry, the neochemotherapy plus liver resection group must be histopathologically diagnosed as ICC before chemotherapy, and the liver resection alone group must be pathologically confirmed as intrahepatic cholangiocarcinoma after surgery;
5. Resectable ICC patients with high risk of LN metastasis (Probability of LN metastasis ≥50% as evaluated by radiomics model);
6. The subject has at least 1 measurable liver disease (according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1);
7. For women who are not breastfeeding or pregnant, use contraception during treatment or 3 months after the end of treatment.
8. The functional indicators of important organs meet the following requirements:

1) Neutrophils≥1.5*109/L; platelets≥90*109/L; hemoglobin≥9g/dl; serum albumin≥3.5g/dl; 2) Coagulation function: International standardization (prothrombin time) ratio (INR) <1.2; 3) Thyroxine (T3 and T4) do not exceed the normal upper and lower limits by 2 times; 4) Bilirubin ≤ 1.5 times the upper limit of normal; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal; 5) Serum creatinine ≤ 1.5 times the upper limit of normal, creatinine clearance ≥ 60ml/min;

Exclusion Criteria:

1. Pathological diagnosis of hepatocellular carcinoma, mixed hepatocellular carcinoma and other non-biliary cell carcinoma malignant tumor components;
2. Patients who have recurrent ICC after surgery, or have chemotherapy in the past;
3. Past or simultaneous suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary carcinoma;
4. Active tuberculosis infection. Patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, no formal anti-tuberculosis treatment or tuberculosis is still active;
5. Suffer from active, known or suspected autoimmune diseases. Subjects with hypothyroidism who only need hormone replacement therapy and skin diseases without systemic therapy can be selected;
6. Past interstitial lung disease, or (non-infectious) pneumonia and need oral or intravenous steroid therapy;
7. Long-term use of systemic hormones (dose equivalent to >10mg prednisone/day) or any other form of immunosuppressive therapy is required. Subjects using inhaled or topical corticosteroids can be selected;
8. Active infections that require systemic treatment;
9. Human immunodeficiency virus (human immunodeficiency virus [HIV], HIV1/2 antibody) positive;
10. A history of psychotropic drug abuse, alcohol or drug abuse;
11. Significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment;
12. Suspected of being allergic to study drugs;
13. Suffer from hypertension, and cannot be well controlled by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
14. After antiviral therapy, hepatitis B virus (HBV)-DNA>104 copies/ml, hepatitis C virus (HCV)-RNA>1000;
15. Accompanied by ascites, hepatic encephalopathy, Gilbert syndrome, sclerosing cholangitis, etc. Combined with insufficiency of other organs, it is expected that they cannot accept general anesthesia or hepatectomy;
16. Other factors judged by the investigator that may affect the safety of the subject or the compliance of the trial. Such as serious illnesses (including mental illness) that require combined treatment, serious laboratory abnormalities, other family or social factors, or participating in other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 24 months
  The time period from randomization to the occurrence of the following events: disease progression prevents liver resection; local or distant recurrence; second primary tumor; death due to various causes.

SECONDARY OUTCOMES:
Overall survival | 36 months
  The time period from the randomization of the patient to the death event due to any reason.
Objective response rate | 4 months
  The proportion of patients whose tumor volume has decreased to a predetermined value.
Adverse events | 6 months
  The severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard the severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard the severity of adverse events will be evaluated according to the NCI CTCAE 5.0 standard.